CLINICAL TRIAL: NCT01355692
Title: Phase III Multi Center Study Study of the Effects of Selective Retinal Photocoagulation for the Treatment of Diabetic Macular Edema
Brief Title: Evaluation of the Effects of Selective Photocoagulation for the Treatment of Diabetic Macular Edema
Acronym: SRT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lumenis Be Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUM.NOVUS SRT.01
Record Dates: First submitted 2011-05-15; First posted 2011-05-18 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Diabetic Macular Edema
Keywords: DME; Laser; Selective laser therapy; photocoagulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Laser therapy (Experimental)
  Interventions: Device: Nd: YLF laser treatment

INTERVENTIONS:
Device: Nd: YLF laser treatment — grid selective retinal treatment
  Other Names: SRT

SUMMARY:
The population of people suffering from diabetes is rapidly increasing, from an estimated 110 million in 1994 to 221 million in 2010. Diabetic macular edema is the most common reason for reduction in visual acuity in diabetic patients.

The standard care for diabetic macular edema is focal and /or grid retinal photocoagulation. During photocoagulation, small laser burns are applied to the retina, the sensory tissue that lines the back of the eye. Studies have shown that photocoagulation of clinically significant diabetic macular edema substantially reduces the risk of visual loss, increase the chance of visual improvement and decrease the frequency of persistent macular edema. However, it remains unknown whether the destruction of sensory layer of the retina during photocoagulation that may cause visual field defects is necessary for successful treatment or is just an unwanted and unnecessary side effect.

Based on these concept, a photocoagulation technique was developed to treat the retina selectively (SRT - Selective retinal therapy), with minimal or no damage to the sensory layers. While the treatment is very similar to regular photocoagulation, the SRT laser uses much lower energy and very short pulses. As a result, treatment does not result in visible burns to the retina and previous studies have shown that the sensory layer remains intact.

The aim of this study is to determine the effect of SRT on the resolution of the edema.

ELIGIBILITY:
Inclusion Criteria:

1. Best corrected ETDRS visual acuity letter score >=24 (app. 20/320 or better)
2. Definite retinal thickness due to diabetic macular edema by on clinical exam at or within 500 to 3000 microns of the macular center (radius) for which the investigator believes laser photocoagulation is not indicated
3. A thickness equal or less than 315 microns in the central subfield (confirmed by SD-OCT).
4. A thickness of >2 SD of norm in one or more inner or outer subfields on SD-OCT.
5. Maximal focal/grid laser not yet applied (within areas of thickening between 500 and 3000 microns from center of macula, not all microaneurysms treated with direct laser and not all other areas of thickening treated with grid laser). Maximal or complete laser treatment is defined as direct treatment to all microaneurysms within areas of edema and grid treatment to all other areas of macular edema.
6. No panretinal scatter photocoagulation (PRP) within prior 4 months.
7. No recent medical treatment for DME (e.g., intravitreal/peribulbar steroids within past 4 months or intravitreal anti-VEGF injection within past 2 months).
8. No major ocular surgery (including cataract extraction, any other intraocular surgery, scleral buckle, glaucoma filter, cornea transplant, etc.) within prior 6 months.
9. No Nd:YAG laser capsulotomy within prior 2 months.
10. Macular edema is not considered to be due to a cause other than diabetic macular edema

    o An eye should not be considered eligible (1) if the macular edema is considered to be related to cataract extraction or (2) clinical exam and/or SD-OCT suggests that vitreoretinal interface disease (eg. vitreoretinal traction or epiretinal membrane) is the primary cause of the macular edema.
11. Media clarity, pupillary dilation, and patient cooperation sufficient for adequate fundus photos.
12. No ocular condition (other than diabetes) that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the first 12 months of the study (e.g., vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, Irvine-Gass Syndrome).

    * Glaucoma per se is not an exclusion

Exclusion Criteria:

1. History of renal failure requiring dialysis or renal transplant
2. Condition that in the opinion of the investigator would preclude participation in the study (e.g., unstable medical status including blood pressure and glycemic control)
3. Patients in poor glycemic control who recently (>3 months) initiated intensive insulin treatment (a pump or multiple daily injections) or plan to do so in the next 3 months should not be enrolled.
4. A patient with only one functioning eye (i.e., letter score 0 in contra-lateral eye)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-12; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
progression of macular edema | 12months
  Proportion progressing to center involved macular edema by month 12 as confirmed on SD-OCT

CONTACTS AND LOCATIONS:
Overall Officials: Anat Loewenstein, MD, Study Director — Tel-Aviv Sourasky Medical Center; Joseph Moisseiev, Prof., Study Director — Sheba Medical Center
Locations (2):
- Israel (2):
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Hahsomer